CLINICAL TRIAL: NCT00390871
Title: Acute Neurological ICU Sedation Trial (ANIST)
Acronym: ANIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANIST
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Sedation
MeSH Terms: interventions — Fentanyl; Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fentanyl/Propofol sedation first (Active Comparator): Patient given fentanyl only first, then sedated with fentanyl/propofol as needed to have Richmond Agitation Sedation Scale (RASS) Score 0 to -1. After washout with fentanyl only, patient sedated with fentanyl/dexmedetomidine to have RASS Score 0 to -1.
  Interventions: Drug: Fentanyl/Dexmedetomidine; Drug: Fentanyl/Propofol; Drug: Fentanyl
- Fentanyl/Dexmedetomidine sedation first (Active Comparator): Patient given fentanyl only first, then sedated with fentanyl/dexmedetomidine as needed to have RASS Score 0 to -1. After washout with fentanyl only, patient sedated with fentanyl/propofol to have RASS Score 0 to -1.
  Interventions: Drug: Fentanyl/Dexmedetomidine; Drug: Fentanyl/Propofol; Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl/Dexmedetomidine
  Other Names: Precedex
Drug: Fentanyl/Propofol
  Other Names: Diprivan
Drug: Fentanyl

SUMMARY:
Dexmedetomidine (Precedex, Hospira) is a "super" selective alpha2-agonist - 8-10x more avid binding to alpha2 receptors than clonidine - and may have particularly favorable characteristics as a continuous i.v. infusion sedative for critically ill neuroscience patients. Its combination of anxiolysis, analgesia, without undue lethargy may make it an ideal agent where frequent neurological examinations are important. Unclear, however, is whether Precedex is superior to current common i.v. sedation protocols, and if there are any undue concerns of this agent on cerebral physiology and cortical stimulation.

DETAILED DESCRIPTION:
Dexmedetomidine has shown promise in small case series to be an efficacious sedative agent in the intensive care unit (ICU) setting, in both post-surgical and medical patients. A recent publication reported on the efficacy in a small series of medical patients (n=12), but as part of the exclusion criteria were any serious nervous system trauma or direct central nervous system (CNS) pathology.

A potential advantage of dexmedetomidine as a sedative agent compared to current popular classes of drugs, particularly propofol, benzodiazepines, and narcotics, is the nominal effect on reduction of level of arousal. Experience suggests that this agent may induce effective degrees of sedation without concomitant loss of attentive behavior and cognition following low levels of auditory or tactile stimulation. Thus, neurological assessment may be preserved while achieving the goal of a non-agitated or anxious patient. Additionally, the combination of both sedative/anxiolytic and analgesic action of dexmedetomidine may permit single drug use for both sedation and pain control during the post-operative and medical ICU period.

The cerebral effects of alpha2-agonists have been modestly studied in the clinical environment, and only in normal volunteers. As expected, cerebral blood flow decreased following initiation of the sedative, coincident with the expected diminishment of global cerebral metabolism. No studies have evaluated dexmedetomidine in patients suffering from neurological injury, the very population that may most benefit from the agent's sedative characteristics. Thus, it is imperative that a safety & efficacy study be carried out in a population of both medical and post-operative neuroscience patients. From an intraoperative perspective, dexmedetomidine has been effectively used as a sedative for both awake and sedation cases. Some evidence suggests prolonged cognitive deficits may persist beyond the sedative action of the drug.

One concern in the neuroscience patient population is laboratory evidence that alpha2-agonists may lower the seizure threshold. Such data has been shown for both clonidine and dexmedetomidine.

Therefore, to provide a comprehensive evaluation leading to successful safety and efficacy data for this sedative, it will be important to perform the following three studies. All three studies will be done concurrently but enrollment between the three studies will be mutually exclusive.

Objective 1: Evaluation of Quality of Sedation: Does dexmedetomidine provide superior sedative characteristics relative to current standard agents in patients with neurological dysfunction? The metrics for such a study will include -

1. Pharmacodynamic ease of sedation: time to goal, required nursing interventions to goal;
2. Quality & consistency of sedation: ability to examine the patient, number of required titration interventions;
3. Rapid weaning: time to off and no residual effect both hemodynamic and neurologic;
4. Systemic hemodynamic alterations requiring drug infusion adjustment or medical intervention;
5. Side effect and toxicity of sedative infusion: neurological dysfunction - cognitive, motor, sensory; electrolyte/hematological/metabolic disturbances, alteration of drug levels.

Objective 2: Alteration of Cerebral Physiology: Does Dexmedetomidine alter intracranial physiology either in a favorable or unfavorable manner? The metrics for such a study will include -

1. Measures of intracranial pressure (ICP), mean arterial pressure (MAP), cerebral perfusion pressure (CPP);
2. Cognitive neurological state;
3. Cerebral saturation (venous) or direct cerebral oximetry (oxygen tissue level) in a subset population with specific intracranial device.

ELIGIBILITY:
Objective 1: Inclusion Criteria:

Neuroscience patients in the Neuro Critical Care Unit (NCCU) who are:

* 18-80 years of age;
* Mechanically ventilated patients;
* Requiring continuous sedation for a minimum of 9-11 hours (depending on whether or not pt is post-operative), yet frequent neurological examinations or Patients with a Nursing Instrument for Communication of Sedation Score (NICSS) > 0
* Patient or family able to provide consent.
* Considered to have guarded yet stable neurological state. Not fluctuating intracranial pressure (ICP), cerebral perfusion pressure (CPP), or ongoing known cerebral ischemia if ICP monitoring in place.

Objective 1: Exclusion Criteria:

* Pregnancy.
* ICP> 30 mm Hg despite therapy if ICP monitored.
* CPP <70 mm Hg if monitored.
* Occurrence of: new cerebral stroke, hemorrhage, or change in edema by CT, increase in ICP if monitored.
* Neuromuscular paralysis.
* Non-functional cognitive exam - not following commands.
* Renal insufficiency: Serum Creatinine >2.0 mg/dl or estimated Cr Clearance <40.0 ml/min.
* Hepatic disease: aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 300, or international normalized ratio (INR) > 1.7 not on anticoagulants.
* Severe chronic obstructive pulmonary disease (COPD) with baseline arterial partial pressure of carbon dioxide (pCO2)>50.
* Suspected alcohol or substance withdrawal.
* Hypotension - requiring pressor therapy to maintain baseline adequate CPP or mean arterial pressure (MAP).
* Cardiac arrhythmia - sinus bradycardia (HR <60), atrial fibrillation (>6 PVC's/min)
* Bradycardia- heart rate less than 60 beats per minute.
* Patient does not require mechanical ventilation.

Objective 2: Inclusion Criteria:

Critically ill neuroscience patients who are:

* 18-80 years of age;
* Mechanically ventilated;
* Require Intracranial Pressure (ICP) monitoring by either subarachnoid bolt (SA bolt), or by an Intra-Ventricular Catheter (IVC).
* Amenable for placement of intra-cerebral oxygen sensor or jugular bulb catheter.
* Have glaucoma coma score (GCS) score > 5 that requires sedation.
* Requiring continuous sedation for minimum of 9-11 hours (depending on whether or not pt is post-operative) , yet frequent neurological examinations every 1-2 hours or Patients with a NICSS score > 0
* Patient or family able to provide consent.

Objective 2: Exclusion Criteria:

* Pregnancy;
* ICP> 30 mm Hg despite therapy; 3) CPP <70 mm Hg;
* Occurrence of: new cerebral stroke, hemorrhage, or change in edema by CT, increase in ICP if monitored.
* Continuous neuromuscular paralysis
* Renal insufficiency: Serum Creatinine >2.0 mg/dl or estimated Cr <40.0 Clearance ml/min.
* Hepatic disease: AST, ALT > 300, or INR > 1.7 not on anticoagulants.
* Severe COPD with baseline arterial pCO2>50.
* Suspected alcohol or substance withdrawal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Johns Hopkins Adapted Cognitive Exam | day of study
  Cognitive assessment tool
Confusion Assessment Method (CAM) for the Intensive Care Unit | day of study
  CAM-ICU delirium assessment tool
Time from initiation of study drug to calm, non-anxious state | day of study
  From control state to RASS Score or 0 to -1 (average=137 min)

SECONDARY OUTCOMES:
Therapy Intensity Level Scale (TIL) | day of study
  Bedside assessment tool to quantify nursing effort
Requirement for fluids, pressors | day of study
  Documenting need for adjunctive treatment with vasoactive agents
Toxicity/side effects | day of study
  documenting drug toxicity - rash, angioedema, nausea, fever, etc.
Numerical Pain Rating Scale | day of study
  behavioral and numerical pain rating
Need for less or more fentanyl during the infusion drug phase | day of study
  assessment of fentanyl dosing required to maintain behavioral pain score at < 3

CONTACTS AND LOCATIONS:
Overall Officials: Marek Mirski, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lewin JJ 3rd, LeDroux SN, Shermock KM, Thompson CB, Goodwin HE, Mirski EA, Gill RS, Mirski MA. Validity and reliability of The Johns Hopkins Adapted Cognitive Exam for critically ill patients. Crit Care Med. 2012 Jan;40(1):139-44. doi: 10.1097/CCM.0b013e31822ef9fc. PMID 21926576